CLINICAL TRIAL: NCT01619189
Title: Thérapie Cellulaire au Cours Des Syndromes d'Insuffisance en Cellules Souches Limbiques
Brief Title: Cell Therapy in Failure Syndromes in Limbal Stem Cells
Acronym: TC181
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Collaborators: Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHRC 2001; AOM01086 (Other: AFSSAPS)
Record Dates: First submitted 2012-05-23; First posted 2012-06-14 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Limbal Deficiency
Keywords: Cell therapy; Limbal deficiency; Limbal stem cell; Transplantation

STUDY DESIGN:
Intervention Model Description: Prospective Phase II Interventional Clinical Trial (Transplantation of Allogeneic or Autologous Limbal Epithelial Stem Cells Cultured on Human Amniotic Membrane with no Feeders)
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tranplantation of cultured LSC in stage 3 limbal deficiency (Experimental): Transplantation of Allogeneic or Autologous Limbal Epithelial Stem Cells Cultured on Human Amniotic Membrane with no Feeders in stage 3 unilateral or bilateral limbal stem cell deficiency.
  Interventions: Biological: epithelial stem cells cultured; Procedure: transplantation of cultured cells

INTERVENTIONS:
Biological: epithelial stem cells cultured — transplantation of allogeneic or autologous limbal epithelial stem cells cultured on human amniotic membrane with no feeders
Procedure: transplantation of cultured cells — transplantation of allogeneic or autologous limbal epithelial stem cells cultured on human amniotic membrane with no feeders

SUMMARY:
Transplantation of allogeneic or autologous limbal epithelial stem cells cultured on human amniotic membrane with no feeders in eyes with total limbal deficiency. Prospective non-comparative monocentric study.

DETAILED DESCRIPTION:
The limbal stem cell deficiency syndrome is characterized by invasion of the corneal surface by an epithelium with a conjunctival differentiation, and, clinically, by opacification and vascularization of the corneal epithelium with impaired corneal epithelial cicatrisation and corneal ulcers that may lead to corneal perforation. When total, the limbal deficiency syndrome is the cause of major disability. Vision decreases largely under the legal threshold of blindness. Overall, the most frequent etiology is by far the complete loss of limbal stem cells induced by severe ocular burns. Until a rather recent date, no treatment was possible in this pathology. Progress in the comprehension of the physiology of the corneal epithelium renewal made it possible to introduce a therapeutic approach, i.e., transplantation of cultured limbal stem cells retrieved from the healthy contralateral eye (autograft, unilateral diseases) or from a cadaveric donor eye (allograft, bilateral diseases or unique eye). Techniques of cell therapy were first described in Italy, Asia and in the USA with positive clinical results. They have all different processes for preparing the cell product to be transplanted and none answers the safety criteria required by the French legislation. The investigators developed a process for preparing a cell therapy product which was accepted by the French regulation agency (AFSSaPS) for a clinical trial (TC181) which began in 2007. The aims of the study are (1) evaluation of the clinical results of this technique in terms of improvement of visual function, reduction in the handicap, improvement of the anatomical condition of the ocular surface and restitution of the physiological function of the limbal epithelium and (2) evaluation of its possible side effects. It is a biphasic monocentric non-comparative prospective study including, according to the clinical responses observed during the first phase (plane of Gehan, ß = 10%), from 15 to 50 voluntary patients with unilateral or bilateral total limbal deficiency. Patient follow-up is 3 years. The expected minimal success rate is 20% for allografts and 40% for the autografts. Monitoring is ensured by URC-Est. The grafts are prepared by culture of autologous or allogeneic limbal epithelial cells from limbal explants on human amniotic membrane. The medical safety requirements relating to transplantation of tissues and cells are reached and the cell therapy products are secured at each stage of their preparation by conventional bacteriological and fungal tests and viral and bacterial PCR. The graft quality is controlled before transplantation. The main outcome measure is survival of the grafted epithelium (Kaplan-Meier method) defined by absence of recurrence of the clinical signs of limbal deficiency (opacification of the corneal epithelium, irregularity of the corneal epithelium, surface corneal vascularization) in the central cornea. The expected repercussions are (1) restitution of a limbal epithelial function allowing a clear corneal epithelium to be obtained, with no superficial vascularization nor chronic epithelial defects, (2) improvement of vision in blind patients, and (3) obtaining a vision higher than the legal threshold of blindness after cell therapy or after subsequent corneal transplantation. If the clinical trial makes it possible to show the effectiveness of this cell therapy technique, a request for authorization of process will be made at AFSSaPS for routine use.

ELIGIBILITY:
Inclusion Criteria:

* Patient age between 18 and 70 years
* Informed consent.
* Unilateral or bilateral limbal deficiency with diffuse opacification of the corneal epithelium, and superficial (or superficial and deep) corneal vascularization, and irregular corneal epithelial surface at slit-lamp examination with fluorescein, either associated with chronic epithelial defects
* Visual acuity of the eye to be treated < 20/20.
* Absence de kératinization of the ocular surface.
* Schirmer test > 0 at 3 minutes.
* For autografts : sérology HIV -, HCV -, HBs

Exclusion Criteria:

* Age < 18 y or > 70 y.
* Absence of informed consent or imformed consent not possible.
* Partial limbal deficiency (healthy corneal epithelium persistant in at least one zone).
* Previous treatment of limbal deficiency by limbal transplantation or amniotic membrane transplantation during the last 12 months.
* Conjunctival stem cell deficiency (xerophtalmia, keratinization of the ocular surface).
* Local anesthesia impossible.
* Immune keratitis not controlled by medical treatment.
* Ocular burn during the last 2 weeks.
* Corneal anesthesia.
* Pregnancy, breast-feeding.
* Allergy to steroid eyedrops.
* Active fungal keratitis.
* For autografts : risk factor for rabbies or Creutzfeldt-Jacob disease, serology HIV +, VHC +, HBs+.
* Follow-up not possible

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2017-03-06 (Actual); Study Completion 2017-03-06 (Actual)

PRIMARY OUTCOMES:
survival of the transplanted epithelium | 3 years
  survival of the transplanted epithelium defined by absence of recurrence of the clinical signs of limbal deficiency (opacification of the corneal epithelium, irregularity of the corneal epithelium, surface corneal vascularization) in the central cornea.

SECONDARY OUTCOMES:
visual acuity | 3 years
  far best spectacle-corrected LogMAR visual acuity
re-epithelialization time after keratoplasty | 3 years
  The healing time of corneal epithelium will be collectively assed by investigators form the CRF and the pictures taken during the study.
Symptoms | 3 years
  Symptoms recorded at each visit:
  * redness : absent (0) - present (1)
  * pain : absent (0) - present (1)
  * burning : absent (0) - present (1)
  * foreign body sensation : absent (0) - present (1)
  * photophobia : absent (0) - present (1)
  * blurred vision : absent (0) - present (1)
  Grading of symptoms : sum of all symptoms (0-6)
morphometric analysis of the ocular surface | 3 years
  the morphometric analysis of the corneal epithelial ulcerations will be assed by the CRA from the pictures of the corneal surface.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent M Borderie, MD, PhD, Principal Investigator — CHNO des 15-20
Locations (1):
- CHNO des quinze-vingts, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borderie VM, Ghoubay D, Georgeon C, Borderie M, de Sousa C, Legendre A, Rouard H. Long-Term Results of Cultured Limbal Stem Cell Versus Limbal Tissue Transplantation in Stage III Limbal Deficiency. Stem Cells Transl Med. 2019 Dec;8(12):1230-1241. doi: 10.1002/sctm.19-0021. Epub 2019 Sep 5. PMID 31486585